CLINICAL TRIAL: NCT03644888
Title: Effects of Continuous Chest Wall Vibration on Dyspnea and Exercise Tolerance in COPD Patients
Brief Title: Continuous Chest Wall Vibration in COPD Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Principal Investigator, Riccardo Buraschi, Principal Investigator, Fondazione Don Carlo Gnocchi Onlus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Vibra_COPD_FDG
Record Dates: First submitted 2018-08-17; First posted 2018-08-23 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: COPD
Keywords: COPD; Vibration; Rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Active Comparator): Cycle ergometer training program: 2 minutes warm-up at no load, 20 minutes at 60% of peak work (PW) calculated by stress-test or at 50% of PW calculated according to Luxton equation (PW = 103.217 + (30.50 X gender) + (-1.613 X age) + (0.002 X 6MWW [m kg -1 ]). The progression of the workloads is calculated according to the BORG Dyspnea and Fatigue Scale (Borg D and F < 5: 10W increase; Borg D and/or F between 5 e 6: maintain same workload; Borg D and / or > 6: 10W decrease) Patient tailored airway clearance program guided by an experienced respiratory physical therapist, which could includes active cycle of breathing technique (ACBT), forced expiratory technique (FET), ELTGOL (slow expiration with glottis open in the lateral position) and PEP techniques (positive expiratory pressure).
  Interventions: Other: Cycle ergometer training; Other: Airway clearance program
- Experimental group (Experimental): Cycle ergometer training program plus application of vibration therapy. The vibration is provided at 150Hz via 4 effectors applied bilaterally at the second or third interspaces in the parasternal region of the upper chest wall and at the seventh to ninth interspaces anterior to the midaxillary line in the lower chest wall.
  Interventions: Other: Cycle ergometer training; Other: Airway clearance program; Device: Vibration therapy
- Sham intervention group (Sham Comparator): Cycle ergometer training program plus application of sham vibration therapy: 4 effectors on chest-wall at same position of vibration therapy, the device that produces vibration is switched on, producing the typical noise and vibration is emitted by effectors not placed on the patient but left in place on the device.
  Interventions: Other: Cycle ergometer training; Other: Airway clearance program; Device: Sham vibration therapy

INTERVENTIONS:
Other: Cycle ergometer training — Already in arm/group descriptions
Other: Airway clearance program — Already in arm/group descriptions
Device: Vibration therapy — Already in arm/group descriptions
  Arms: Experimental group
Device: Sham vibration therapy — Already in arm/group descriptions
  Arms: Sham intervention group

SUMMARY:
Dyspnea, the sensation of breathing discomfort or shortness of breath, is one of the main symptoms for patients affected by Chronic Obstructive Pulmonary Disease (COPD), particularly during exercise. Previous study show that chest wall vibration decrease dyspnea in COPD patients and precisely when applied during the inspiration phase, called "in-phase vibration" (IPV) which provide vibration directly on intercostal muscles. These findings have been obtained in laboratory context and the intercostals muscles vibration has been tested only in single phases of breathing, during inspiration with IPV and during exhalation with out-of-phase vibration (OPV). None study has evaluated the effect of a continuous chest wall vibration (CCWV), namely muscles vibration during the whole cycle of breathing, on dyspnea in patients with COPD in a clinical context. Continuous high frequency vibration has been proven to reduce myoelectrical manifestation of fatigue, probably modifying the centrally driven motor unit recruitment hierarchy, in healthy subjects.

Moreover, CCWV is a modality of provide vibration more suitable and cost-effective in a clinical context than single-phases vibration that requires specific instruments for the detection of breathing phases and the coupling with vibration device.

On these bases, the investigators hypothesized that CCWV at high frequency, applied during a cycle ergometer training program, could decrease dyspnea and enhance the exercise tolerance in COPD patients. Therefore, the aim of this study is to evaluate the effects of high frequency CCWV on dyspnea and exercise tolerance in patients with COPD patients compared to usual care and to sham intervention.

ELIGIBILITY:
Inclusion Criteria:

- COPD diagnosis (GOLD stage: 2-3-4)

Exclusion Criteria:

* Restrictive lung disease
* Active pulmonary infection
* Pulmonary embolism (less than 3 months)
* Pneumotorax
* Thoracic/abdominal operation (less than 3 months)
* Myocardial infarction (less than 6 months)
* Congestive heart failure/ heart failure/ right heart failure
* Angina/severe angina
* Incapability of perform the cycle ergometer training (e.g. orthopaedic or urogenital conditions)
* Incapability to understand the intructions required to carry out the tests and assessments planned

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-09-12 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Change of Dyspnea | Change from Baseline Barthel Index based on dyspnea at 4 weeks
  Barthel Index based on dyspnea. The scale measures the level of dyspnea perceived in performing basic daily living activities, Range: 0 - 100 Higher values represent a worse outcome
Change of exercise tolerance | Change from Baseline exercise tolerance at 4 weeks
  Six Minutes Walking Test. This test assesses distance walked over 6 minutes as a sub-maximal test of aerobic capacity/endurance.
  Higher values represent a better outcome

SECONDARY OUTCOMES:
Change of respiratory muscles strength | Change from Baseline respiratory muscles strength at 4 weeks
  Maximum inspiratory pressure / Minimum expiratory pressure.
  Maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP) are global measures of maximal strength of respiratory muscles and they are respectively the greater pressure which may be generated during maximal inspiration and expiration against an occluded airway. The way to measure maximal respiratory pressures is very simple, using a hand-held mouth pressure meter in cmH2O.
  Higher values represent a better outcome
Change of Risk of death | Change from Baseline risk of death at 4 weeks
  BODE Index.
  Is a multidimensional 10-point grading system that predicts the risk of death from any cause and from respiratory causes among patients with COPD. It is composed by subscales, combined to compute a total score as follows:
  FEV1 (% of predicted): 0 (≥65); 1 (50-64); 2 (36-49); 3 (≤35). Distance walked in 6 minutes (m): 0 (≥350); 1 (250-349); 2 150-249); 3 (≤149). MMRC dyspnea scale:0 (0-1); 1 (2); 2 (3); 3 (4). Body-mass Index: 0 (>21); 1 (≤21).
  Range: 0-10 Higher scores indicate a worse outcome (higher risk of death)
Change of Health-related quality of life | Change from Baseline health-related quality at 4 weeks
  Saint George Respiratory Questionnaire. Is a self-reported, disease-specific, health-related quality of life questionnaire.
  Range: 0 (no health impairment) - 100 (maximum health impairment).
  Higher values represent a worse outcome
Change of Sympatho-vagal balance | Change from Baseline sympatho-vagal balance at 2 weeks and at 4 weeks
  Heart Rate Variability

CONTACTS AND LOCATIONS:
Overall Officials: Riccardo Buraschi, DPT, Principal Investigator — IRCCS Fondazione Don Carlo Gnocchi
Locations (1):
- Fondazione Don Carlo Gnocchi Onlus - Centro Ettore Spalenza, Rovato, Brescia, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Binks AP, Bloch-Salisbury E, Banzett RB, Schwartzstein RM. Oscillation of the lung by chest-wall vibration. Respir Physiol. 2001 Jul;126(3):245-9. doi: 10.1016/s0034-5687(01)00223-7. PMID 11403786
- [Background] Bolser DC, Lindsey BG, Shannon R. Respiratory pattern changes produced by intercostal muscle/rib vibration. J Appl Physiol (1985). 1988 Jun;64(6):2458-62. doi: 10.1152/jappl.1988.64.6.2458. PMID 3403429
- [Background] Burke D, Hagbarth KE, Lofstedt L, Wallin BG. The responses of human muscle spindle endings to vibration during isometric contraction. J Physiol. 1976 Oct;261(3):695-711. doi: 10.1113/jphysiol.1976.sp011581. PMID 135841
- [Background] Cardinale M, Bosco C. The use of vibration as an exercise intervention. Exerc Sport Sci Rev. 2003 Jan;31(1):3-7. doi: 10.1097/00003677-200301000-00002. PMID 12562163
- [Background] Cristiano LM, Schwartzstein RM. Effect of chest wall vibration on dyspnea during hypercapnia and exercise in chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 1997 May;155(5):1552-9. doi: 10.1164/ajrccm.155.5.9154856.
- [Background] Fallon JB, Macefield VG. Vibration sensitivity of human muscle spindles and Golgi tendon organs. Muscle Nerve. 2007 Jul;36(1):21-9. doi: 10.1002/mus.20796. PMID 17471568
- [Background] Casale R, Ring H, Rainoldi A. High frequency vibration conditioning stimulation centrally reduces myoelectrical manifestation of fatigue in healthy subjects. J Electromyogr Kinesiol. 2009 Oct;19(5):998-1004. doi: 10.1016/j.jelekin.2008.08.002. Epub 2008 Sep 26. PMID 18819821
- [Background] Nakayama H, Shibuya M, Kaneko N, Yamada M, Suzuki H, Arakawa M, Homma I. Benefit of in-phase chest wall vibration on the pulmonary hemodynamics in patients with chronic obstructive pulmonary disease. Respirology. 1998 Dec;3(4):235-40. doi: 10.1111/j.1440-1843.1998.tb00128.x. PMID 10201049
- [Background] Nakayama H, Shibuya M, Yamada M, Suzuki H, Arakawa M, Homma I. In-phase chest wall vibration decreases dyspnea during arm elevation in chronic obstructive pulmonary disease patients. Intern Med. 1998 Oct;37(10):831-5. doi: 10.2169/internalmedicine.37.831. PMID 9840703
- [Background] Sibuya M, Yamada M, Kanamaru A, Tanaka K, Suzuki H, Noguchi E, Altose MD, Homma I. Effect of chest wall vibration on dyspnea in patients with chronic respiratory disease. Am J Respir Crit Care Med. 1994 May;149(5):1235-40. doi: 10.1164/ajrccm.149.5.8173764.
- [Background] Bausewein C, Booth S, Gysels M, Higginson I. Non-pharmacological interventions for breathlessness in advanced stages of malignant and non-malignant diseases. Cochrane Database Syst Rev. 2008 Apr 16;(2):CD005623. doi: 10.1002/14651858.CD005623.pub2. PMID 18425927
- [Derived] Pancera S, Buraschi R, Bianchi LNC, Porta R, Negrini S, Arienti C. Effectiveness of Continuous Chest Wall Vibration With Concurrent Aerobic Training on Dyspnea and Functional Exercise Capacity in Patients With Chronic Obstructive Pulmonary Disease: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2021 Aug;102(8):1457-1464. doi: 10.1016/j.apmr.2021.03.006. Epub 2021 Mar 26. PMID 33781780